CLINICAL TRIAL: NCT05790317
Title: Comparıson Of The Effects Of The Eras Protocol Applıcatıon And The Effects Of The Tradıtıonal Method On The In Obesıty Surgery
Brief Title: Comparison of the Effect of Traditional Method and Eras Protocol in Obesity Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Eylul Tulay Aykul, training nurse, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Bau-bahcesehir university
Record Dates: First submitted 2022-12-18; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Obesity, Morbid; Bariatric Surgery Candidate; Obesity Adult Onset; Obesity Associated Disorder; Diabetes; Nausea; Ache; Pain, Postoperative; Postoperative Nausea; Postoperative Nausea and Vomiting; Post Procedural Discharge; ERAS; DVT
Keywords: DVT; BKÖİ; DSÖ; ASA; BKI; BPD; CVI; DMAH; ERAS; FTS; IASMEN; MBT; LSG
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus; Nausea; Pain; Pain, Postoperative; Postoperative Nausea and Vomiting | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical Procedure with ERAS Protocol (Experimental): ERAS Maintenance Protocol The basic philosophy of the ERAS Protocol is to reduce metabolic stress due to surgical trauma, and to return to normal activity as soon as possible by supporting the normalization of functions in a short time. ERAS protocols are a protocol consisting of a total of 24 items covering the perioperative period of a patient, which starts in the outpatient clinic in the preoperative period and ends at home with discharge. includes applications. Elements of this preparation and treatment method, which is different from the traditional, were applied to our patients in this group before (11), during the operation (6) and after the operation (7). In the study, the data were collected with the personal introduction form introducing the characteristics of the patients, the Rhodes Nausea-Vomiting and Regurgitation Index (WPI), the Mcgill Pain Scale and the Postoperative Evaluation Form created within the scope of the ERAS Care Protocol.
  Interventions: Procedure: Surgical Procedure with ERAS Protocol
- Surgery Procedure with the traditional method (No Intervention): ItThe group that underwent surgery with the traditional method is the control group. The surgical procedure preparation procedure in the institution where the study was conducted was not exceeded.
  The data in the control group were collected with the patient information form, the Postoperative Evaluation Form to evaluate the symptoms after the surgical intervention, the McGill Pain Scale Short Form, the Rhodes Nausea-Vomiting Regurgitation Index.

INTERVENTIONS:
Procedure: Surgical Procedure with ERAS Protocol — It covers the period before, during and after the surgery.
  Other Names: Fast Track Surgery
  Arms: Surgical Procedure with ERAS Protocol

SUMMARY:
This study was conducted to compare the effectiveness of care based on the "Accelerated Recovery After Surgery (ERAS) Protocol" and the traditional method in bariatric surgery and demonstrate the difference the two methods based on evidence.

DETAILED DESCRIPTION:
The population of the study consisted of 700 patients over the age of 18 who underwent bariatric surgery in the Obesity Surgery Clinic of a private hospital in 2022. The sample of the study included 128 patients who were willing to undergo bariatric surgery between April 15-July 31, 2022, were in compliance with the research criteria and were voluntarily over the age of 18, 64 in the control and 64 in the experimental group. 128 patients in the sample were assigned to 2 groups using a computer program that generates random numbers. For the purpose of the research, groups were coded as groups A and B, and two different surgical preparations and surgical procedures were applied to the patients in the group. The effects of two different surgical method preparations and the surgical process on the patient's recovery were compared. In the study, the data were collected with the personal introduction form introducing the characteristics of the patients, the Rhodes Nausea-Vomiting and Regurgitation Index (WPI), the Mcgill Pain Scale and the Postoperative Evaluation Form created within the scope of the ERAS Accelerated Care Protocol. Permission was obtained for the scales, and the content validity calculation of the Postoperative Evaluation Form was made in line with the evaluations of the field experts consisting of physicians and nurses experienced in the ERAS Rapid Care Protocol. The data were analyzed in SPSS Package Program. While calculating frequency, percentage and standard deviation in the evaluation of the data, comparisons between groups were made with the independent sample t-test, and p≤ 0.05 was taken as the significance value of the findings.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age who underwent bariatric surgery
* Open to communication and collaborative,
* Patients who volunteered to take part in the study

Exclusion Criteria:

* Patients with major visual, hearing and speech impairments
* Patients who want to withdraw from the study at any stage of the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Presence and level of postoperative pain | 3 days
  In the sample calculation of the research; To measure the significant differences between independent groups, a minimum of 128 samples is required (64 for each group) in order to determine 80% statistical power and α = 0.05 significance and d = 0.50 effect size in the t-test to be performed.
  In order to evaluate the effect of the post-operative accelerated recovery (ERAS) protocol on the patient recovery process, 128 patients who applied to the hospital for bariatric surgery between April and June 2022 were included in the study. 64 patients were divided into groups as the ERAS Protocol group and 64 patients as the control group.
  Postoperative pain status was evaluated with the McGill Pain Questionnaire (SF-MPQ). In determining the severity of pain, the McGill Pain Scale Numerical Evaluation was evaluated as 0-10 points, 0 no pain, 10 unbearable pain. A score of 4 or less for patients meant less pain.
Presence of post-operative nausea, vomiting and retching | 3 days
  Postoperative nausea, vomiting and retching were evaluated with the "Rhodes Nausea-Vomiting Rectal Index". According to the sub-dimensions of the scale, each of the symptoms of nausea, vomiting and retching was scored in the range of 0-12 points. 0 meant the least distress - 12 meant the most distress.

CONTACTS AND LOCATIONS:
Overall Officials: Eylül Tülay Aykul, master, Principal Investigator — Bahçeşehir University
Locations (1):
- Bahcesehir university, Istanbul, Besiktas, Turkey (Türkiye)